CLINICAL TRIAL: NCT05882370
Title: TIPS Plus Cadonilimab (a PD-1/CTLA-4 Bispecific Antibody) in Advanced Hepatocellular Carcinoma with Tumor Thrombosis-associated Portal Hypertension: a Prospective, Single-arm, Phase II Study
Brief Title: TIPS Plus Cadonilimab in Advanced HCC with Tumor Thrombosis-associated Portal Hypertension:a Prospective, Single-arm, Phase II Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fei Gao (Other)
Responsible Party: Sponsor-Investigator, Fei Gao, Clinical Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCALE
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: TIPS; Cadonilimab; Combination therapy; advanced HCC; tumor thrombosis-associated portal hypertension
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SCALE (Experimental): TIPS plus Cadonilimab
  Interventions: Drug: Cadonilimab; Procedure: transjugular intrahepatic portosystemic shunt (TIPS)

INTERVENTIONS:
Drug: Cadonilimab — Patients were treated with TIPS plus Cadonilimab (10mg/kg, intravenously, d1, Q3W) to a maximum total cycle of 18 unless any evidence of disease progression or unacceptable side effects.
Procedure: transjugular intrahepatic portosystemic shunt (TIPS) — transjugular intrahepatic portosystemic shunt (TIPS)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of transjugular intrahepatic portosystemic shunt (TIPS) plus Cadonilimab (a PD-1/CTLA-4 bispecific antibody) in advanced hepatocellular carcinoma (BCLC-C Stage) accompanied by tumor thrombosis-associated portal hypertension.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II study to evaluate the efficacy and safety of transjugular intrahepatic portosystemic shunt (TIPS) plus Cadonilimab (a PD-1/CTLA-4 bispecific antibody) in advanced hepatocellular carcinoma (BCLC-C Stage) accompanied by tumor thrombosis-associated portal hypertension. Subjects who meet the admission criteria will be treated with Cadonilimab after TIPS until disease progression, intolerable toxicity, death, withdrawal of the patient, or the researchers determined that the drug must be discontinued.

The primary outcome measure is to evaluate the objective response rate (ORR). The secondary outcome measures include the duration of response (DOR), disease control rate (DCR), overall survival rate (OSR) in 6- and 12-months, the median progression-free survival time (mPFS) and median overall survival time (mOS). This study also aims to assess the safety and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined the study and signed an informed consent form;
2. ≥18 and ≤ 75 years old, both male and female;
3. Clinically diagnosed or pathologically confirmed hepatocellular carcinoma, at least one measurable focus without local treatment (according to mRECIST requirements, the measurable focus spiral CT scan length ≥ 10 mm or enlargement Short diameter of lymph node ≥15 mm);
4. Child-Pugh score ≤ 13 points;
5. BCLC-C stage accompanied by tumor thrombosis-associated portal hypertension;
6. Newly diagnosed patients who have not received targeted therapy or immunotherapy in the past;
7. ECOG score: 0～1;
8. Expected survival period ≥ 12 weeks;
9. The functions of vital organs meet the following requirements (no blood components, cell growth factors and other corrective treatment drugs are allowed within 14 days before the first administration):
10. The absolute count of neutrophils≥1.5×109/L; Platelet ≥50×109/L; Hemoglobin ≥60 g/L; Serum albumin ≥28 g/L; Thyroid-stimulating hormone (TSH)≤1×ULN (if abnormal, the levels of FT3 and FT4 should be examined at the same time, if the levels of FT3 and FT4 are normal, they can be included in the group); Bilirubin≤2×ULN (within 7 days before the first administration); ALT and AST ≤5×ULN (within 7 days before the first dose); Serum creatinine≤1.5×ULN;
11. Non-surgical sterilization or female patients of childbearing age need to use a medically approved contraceptive method (such as an intrauterine device, contraceptive, or condom) during the study treatment period and within 3 months after the end of the study treatment period; Female patients of childbearing age who undergo surgical sterilization must be negative in serum or urine HCG within 72 hours before enrollment in the study; and must be non-lactating; for male patients whose partners are women of childbearing age, at the last time use effective methods for contraception within 3 months.

Exclusion Criteria:

1. The patient has any active autoimmune disease or a history of autoimmune disease;
2. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose>10mg/day prednisone or other curative hormones), and continues to use it within 2 weeks before enrollment;
3. The number of system treatment lines ≥ 2 lines;
4. Severe allergic reaction to other monoclonal antibodies;
5. Those with a known history of central nervous system metastasis or hepatic encephalopathy;
6. Patients who have received liver transplantation in the past;
7. Tumor thrombus beyond the portal vein range, such as hepatic vein, inferior vena cava, right atrium, splenic vein, superior mesenteric vein cancer thrombus, etc.;
8. Suffer from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
9. Uncontrolled cardiac clinical symptoms or diseases, such as: NYHA level 2 or higher heart failure, unstable angina pectoris, myocardial infarction occurred within 1 year, clinically significant supraventricular or ventricular arrhythmia requires treatment or intervention , QTc>450ms (male); QTc>470ms (female);
10. Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow the preventive use of low-dose aspirin and low molecular heparin;
11. Child-Pugh score >13 points;
12. Arterial/venous thrombosis events that occurred within 6 months before randomization, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
13. Known genetic or acquired bleeding and thrombotic tendency (such as hemophilia patients, coagulation dysfunction, thrombocytopenia, etc.); Urine routine test showed urine protein ≥ ++ and confirmed 24-hour urine protein content> 1.0 g;
14. Patients who have previously received radiotherapy, chemotherapy, hormone therapy, and surgery, after the completion of the treatment (last medication) and less than 4 weeks before the study medication; molecular targeted therapy (including other oral targeted drugs used in clinical trials) is less than the first study medication <5 drug half-lives, or patients whose adverse events (except alopecia) caused by previous treatment have not recovered to ≤ CTCAE level 1;
15. The patient has active infection, fever of unknown origin within 7 days before medication ≥38.5℃, or baseline white blood cell count >15×109/L; Patients with congenital or acquired immune deficiencies (such as HIV-infected persons);
16. Moderate to severe pulmonary hypertension, pulmonary artery pressure was assessed by ultrasound >40mmHg；
17. The patient suffered from other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ);
18. Central nervous system metastasis；
19. The patient has previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or has previously received apatinib therapy;
20. Live vaccine may be vaccinated less than 4 weeks before study medication or may be administered during the study period;
21. According to the judgment of the investigator, the patient has other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, and serious laboratory tests 22. Abnormalities, accompanied by family or social factors, will affect the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) by RECIST 1.1 and mRECIST | From date of first dose of study drug until disease progression, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to 2 years)
  ORR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST

SECONDARY OUTCOMES:
Disease control rate (DCR) | From date of first dose of study drug until disease progression, stable disease, development of unacceptable toxicity, withdrawal of consent, or sponsor termination (up to 2 years)
  DCR is defined as the percentage of participants who have best overall response (BOR) of complete response (CR) or partial response (PR) or stable disease (SD) at the time of data cutoff as assessed by RECIST 1.1 and mRECIST.
Duration of response (DOR) | From the first documentation of CR or PR to the first date of documentation of disease progression or death whichever occurs first (up to 2 years)
  DOR is defined as the time from the first documentation of CR or PR to the date of first documentation of disease progression or death (whichever occurs first) as assessed by RECIST 1.1 and mRECIST
Overall survival rate (OSR) | From date of first dose of study drug to the date of first documentation of death from any cause, whichever occurs first (up to 2 years)
  OSR in 6- and 12-months
Progression-free survival time (mPFS) | From date of first dose of study drug to the date of first documentation of disease progression (up to 2 years)
  The progression-free survival time (mPFS) defined as the time from the first study dose date to the date of first documentation of disease progression as assessed by RECIST 1.1 and mRECIST.
Median overall survival time (mOS) | From the start date of the Treatment Phase until date of death from any cause (up to 2 years)
  OS is measured from the start date of the Treatment Phase (date of first study dose) until date of death from any cause. Participants who are lost to follow-up and the participants who are alive at the date of data cutoff will be censored at the date the participant was last known alive or the cut-off date, whichever comes earlier.

OTHER OUTCOMES:
Treatment-related adverse events | From the start date of the Treatment Phase until date of death from any cause (up to 2 years)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China